CLINICAL TRIAL: NCT01073527
Title: Interventional Study: Hypertonic Saline as Add on Treatment to the Usual Therapy for Preschool Children With Acute "Asthmatic" Attack Presenting to the ER: A Double Blind Control Study
Brief Title: Hypertonic Saline as Add on Therapy in Preschool Children With Acute Wheezing Attack.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Avigdor Mandelberg MD, Director, Pediatric Pulmonary Unit, Wolfson Medical Center, Holon, Israel, The Sackler School of Medicine, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1038
Record Dates: First submitted 2009-08-18; First posted 2010-02-23 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2011-08

CONDITIONS: Asthma
Keywords: Child, preschool; Pediatric emergency department
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypertonic saline-salbutamol combination (Active Comparator): NaCl 5% - 4cc (with standard treatment - salbutamol 0.5cc)
  Interventions: Drug: hypertonic saline-salbutamol combination
- normal saline-salbutamol combination (Placebo Comparator): Standard treatment normal saline 4cc with salbutamol 0.5cc
  Interventions: Drug: Normal saline-salbutamol combination

INTERVENTIONS:
Drug: hypertonic saline-salbutamol combination — hypertonic saline 5% with 0.5cc salbutamol
  Other Names: Preschool asthma,Induced sputum, Metacholine,Adenosine
  Arms: Hypertonic saline-salbutamol combination
Drug: Normal saline-salbutamol combination — normal saline - 4cc with salbutamol 0.5cc
  Other Names: Preschool asthma
  Arms: normal saline-salbutamol combination

SUMMARY:
To investigate the efficacy of adding Inhaled Hypertonic Saline treatment (HS) for 1-6 year old children with "asthmatic" attack presenting to Emergency Department (ED).

Background: In 1-6 year old children, the most common causes of acute exacerbations of asthma requiring urgent medical care are viral respiratory infections. Most of these children are not atopic and often do not respond very well to bronchodilators and steroids. Thus novel treatments are needed.

HS is considered an effective and safe treatment for infants with acute viral bronchiolitis (Cochrane 2008). HS acts in the airways in several mechanisms: HS re-hydrates secretions and improving mucus rheology, reduce edema of the airway wall by absorbing water from the mucosa and submucosa, causes sputum induction and cough, which can help to clear the sputum out of the bronchi, stimulates cilial beat via the release of prostaglandin E2, breaks the ionic bonds within the mucus gel, thereby lowering the viscosity and elasticity of the mucus secretion.

It is estimated that all the above HS responding elements may play a role in this viral induce wheezing. The above mentioned theoretical benefits provide the rationale for the possible treatment of viral induced acute wheezing ("asthma") attack with nebulized HS in young pre-school children presenting to the Pediatric Emergency Unit with acute (mostly viral induced) wheezing.

Therefore, the purpose of the present study is to 1. Investigate the addition of frequently nebulized 5% HS/albuterol combination to standard therapy of acute asthmatic episodes presenting to the emergency department (ED) in preschool children in a prospective, randomized, double-blind, controlled fashion.

DETAILED DESCRIPTION:
A randomized double blind, controlled, (DBCR) trial. To investigate the efficacy of adding inhaled Hypertonic Saline (HS) treatment for 1-6 year old children with asthmatic attack presenting to ED

Background:

Children under the age of 5 years have the highest hospitalization rate of asthma. The most common causes of acute exacerbations of asthma requiring urgent medical care are viral respiratory infections. Most of these children < 6 years old are not atopic.

These investigators have previously demonstrated in wheezy infants with acute viral bronchiolitis that nebulized hypertonic saline produces a clinical significant reduction in length of hospital stay and improves the clinical score and is considered an effective and safe treatment for infants with acute viral bronchiolitis (Cochrane 2008).

Hypertonic saline solution acts in the airways in several mechanisms:

It Stimulates ciliar beat via the release of prostaglandin E2 and increases mucociliary clearance.

It Breaks the ionic bonds within the mucus gel, thereby reducing the degree of cross linking and entanglements and lowering the viscosity and elasticity of the mucus secretion.

HS induces an osmotic flow of water into the mucus layer, re-hydrating secretions and improving mucus rheology.

HS reduces edema of the airway wall by absorbing water from the mucosa and submucosa.

HS can cause sputum induction and cough, which can help to clear the sputum outside of the bronchi and thus improve airway obstruction.

It is estimated that many of the above hypertonic saline responding elements may play a role in this viral induce wheezing such as: mucosal and submucosal edema, peribronchial infiltrate of inflammatory cells, necrosis and desquamation of ciliated epithelial cells, and excess mucus secretion. The combination of an airway wall swelling, sloughing of necrotic debris, increased mucus production and impaired secretion clearance, eventually contribute in addition to bronchospasm to airway obstruction, gas trapping, atelectasis and impaired gas exchange. Moreover, as postulated in "status asthmatic", the relative contribution of these "non-spasmodic" pathological and pathophysiological consequences of viral and asthmatic inflammation to airway obstruction, gas trapping, atelectasis and impaired gas exchange become even more important in these children already treated with maximum dilatation dose of bronchodilating drugs in the emergency department.

The above mentioned theoretical benefits provide the rationale for the possible treatment of viral induced acute wheezing ("asthma") attack with nebulized hypertonic saline solution in young pre-school children presenting to the Pediatric Emergency Unit with acute (mostly viral induced) wheezing.

Therefore, the purpose of the present study is to investigate the addition of frequently nebulized 5% HS/albuterol combination to standard therapy of acute asthmatic episodes presenting to the ED in preschool children in a prospective, randomized, double-blind, controlled fashion.

ELIGIBILITY:
Inclusion Criteria:

* Children, age: 1-6 years old
* Presenting to the ED with acute wheezing episode

Exclusion Criteria:

* Any chronic (lung, cardiac, immunologic, neurologic) disease

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2009-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
shortening length of stay (LOS) | From admision to ready to discharge.

SECONDARY OUTCOMES:
Hospitalization rate | From presenting to ED until admission to hospital
Improvement in clinical score (CS) | Post inhalations on presentation to the ED and daily during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Avigdor Mandelberg, MD, Principal Investigator — The Sackler School of Medicine, Tel Aviv University, Israel
Locations (1):
- The Edith Wolfson MC, Holon, Israel

REFERENCES:
- [Derived] Ater D, Shai H, Bar BE, Fireman N, Tasher D, Dalal I, Ballin A, Mandelberg A. Hypertonic saline and acute wheezing in preschool children. Pediatrics. 2012 Jun;129(6):e1397-403. doi: 10.1542/peds.2011-3376. Epub 2012 May 21. PMID 22614767